CLINICAL TRIAL: NCT04733664
Title: A Pilot, Open-Label Study to Evaluate the Safety, Tolerability, and Performance of the FAST PV Technology™ in Chronic Dialysis Patients With Extremely Reduced or No Kidney Function
Brief Title: Pilot Study to Evaluate Safety, Tolerability, and Performance of the FAST PV Technology™ in Chronic Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FAST BioMedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008193898
Record Dates: First submitted 2020-09-01; First posted 2021-02-02 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Cohort 1 (Experimental): Patients will receive one dose of visible fluorescent injectate (VFI)™ and one dose of iohexol approximately 4 hours prior to undergoing dialysis followed by a second dose of VFI and iohexol approximately 1 hour after completing dialysis.
  Interventions: Device: VFI using the FAST PV Technology

INTERVENTIONS:
Device: VFI using the FAST PV Technology — The bolus IV administered visible fluorescent injectate (VFI) agent is comprised of a mixture of 2 different molecular weight carboxymethyl dextran molecules (5 kD and 150 kD) with different fluorescent dye molecules attached.

SUMMARY:
The FAST Plasma Volume (PV) Technology will aid in determining the plasma and interstitial volumes of end stage renal disease patients before and after dialysis therapy, providing a more precise understanding of pre and post dialysis volumes and extent of volume removal during the course of treatment.

DETAILED DESCRIPTION:
This is a pilot, single site, open-label study designed to evaluate the safety, tolerability, and performance of the FAST plasma volume (PV) Technology in dialysis patients.

Administration of VFI will occur within 28 days of screening.

Patients will receive 1 dose of VFI and 1 dose of iohexol approximately 4 hours prior to undergoing dialysis followed by a second dose of visible fluorescent injectate (VFI) and iohexol approximately 1 hour after completing dialysis. Patients will be discharged following completion of Day 1 activities. Patients will be seen and evaluated on their next 2 dialysis sessions for any adverse reaction by answering questions about their health, approximately on Day 3 and Day 8. A follow-up phone call will be performed on Day 31 (± 1 day).

ELIGIBILITY:
Inclusion Criteria:

Subjects/patients must meet all inclusion criteria to be eligible for study participation.

1. Males or females ≥ 18 years of age.
2. Females must be of non-childbearing potential (eg, postmenopausal [defined cessation of regular menstrual periods for at least 1 year confirmed by age => 60 or surgically sterile by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation [documentation required]) or be using a medically acceptable form of birth control (a barrier method, intrauterine device, or hormonal contraception) from screening through 30 days after administration of the last dose of VFI.
3. Males who are sexually active and whose partners are females of childbearing potential must agree to practice abstinence or use condoms from screening through 90 days after administration of the last dose of VFI, and their partners must be willing to use a medically acceptable method of contraception (a barrier method, intrauterine device, or hormonal contraception) from screening through 90 days after administration of the last dose of VFI.
4. Males must agree to not donate sperm from screening through 90 days after administration of the last dose of VFI.
5. Subjects/patients must be able to communicate effectively with the study personnel.
6. Patients must be on chronic hemodialysis for >= 3 months and oliguric defined as <= 2 urinary voids per day.
7. Patients must have an average interdialytic weight gain of at least 2 kg.
8. Patients must have an A-V dialysis shunt.
9. Patients must have a functioning A-V dialysis shunt, either fistula or graft.

Exclusion Criteria Subjects/patients will not be eligible for study participation if they meet any of the exclusion criteria, or will be discontinued at the discretion of the investigator if they develop any of the exclusion criteria during the study.

1. Subject is a pregnant or nursing (lactating) woman, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
2. History or presence of conditions which, in the judgment of the investigator, are known to interfere with the distribution, metabolism, or excretion of drugs
3. History or presence of conditions that may place the subject/patient at increased risk as determined by the investigator.
4. History of surgery or major trauma within 12 weeks of screening or surgery planned within 4 weeks of the study, including during study participation.
5. Has taken other investigational drugs within 30 days or 5 half-lives of the investigational drug's PK, PD, or biological activity, whichever is longer, prior to first dose of VFI in this study.
6. Prior exposure to VFI or known allergy or hypersensitivity to dextran, 5-aminofluorescein dye, or 2-sulfohexamine rhodamine dye.
7. History of any clinically significant allergic or negative reactions, side effects, or anaphylaxis to iodine, dyes, shellfish, isotopes, or dextran molecules.
8. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 4 weeks prior to study participation.
9. Presence of significant hemodynamic instabilities defined as systolic BP <100 on dialysis requiring saline infusion in the past 4 weeks.
10. Presence of ascites and/or 4+ anasarca.
11. Any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.
12. Involved in the planning or conduct of this study.
13. Unwilling or unlikely to comply with the requirements of the study.
14. Clinically significant ongoing bleeding, changing hemoglobin, or experienced significant blood loss within the last 4 weeks.
15. Had a PRBC transfusion in the prior 2 weeks
16. Use of midodrine.
17. Any other condition or prior therapy that, in the investigator's opinion, is likely to deteriorate during study participation
18. Subjects suffering from significant non-cardiac diseases of other organ systems (e. g. Malignancies, significant neurological diseases).
19. Subject has a psychiatric disease or a history of illicit drug use that would prohibit them from complying with study requirements.
20. Use of hemodialysis catheter as primary vascular access for hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Median (Standard Deviation); unit: years] | 58.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Plasma Volume (PV) and Interstitial Volume (ISV) Using the FAST PV Technology and Iohexol in Patients on Chronic Dialysis Pre-dialysis
Description: To measure quantitatively the ISV and PV of patients pre dialysis using the FAST PV Technology and iohexol measurement
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 10
mL
  FAST PV | 3869 (805)
  FAST ISV | 9152 (1701)
  Iohexol PV | 3895 (801)
  Iohexol ISV | 19057 (3376)

2. Primary Outcome: Evaluate Plasma Volume (PV) and Interstitial Volume (ISV) Using the FAST PV Technology and Iohexol in Patients on Chronic Dialysis Post-dialysis
Description: To measure quantitatively the ISV and PV of patients post dialysis using FAST PV Technology and the iohexol measurement
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
mL
  FAST PV | 3615 (963)
  FAST ISV | 7078 (1816)
  Iohexol PV | 3684 (954)
  Iohexol ISV | 16770 (4409)

3. Primary Outcome: Evaluate the Difference in ISV and PV Pre- and Post Dialysis by the FAST PV Technology
Description: Directly compare quantitative difference of ISV and PV measured by the FAST PV Technology to the volume removed during dialysis
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
mL
  FAST PV Difference | 343 (376)
  FAST ISV Difference | 2284 (680)
  FAST Total Volume Removed | 2628 (904)
  Total Volume removed as measured by UF | 2451 (604)

4. Primary Outcome: Evaluate the Difference of ISV and PV Pre- and Post Dialysis by Iohexol
Description: Directly compare quantitative difference of ISV and PV measured by the Iohexol measurement to the volume removed during dialysis
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1
Number analyzed (Participants) | 9
mL
  Iohexol PV Difference | 340 (380)
  Iohexol ISV Difference | 2537 (2012)
  Iohexol Total Volume Removed | 2877 (1940)
  Total Volume removed measured by UF | 2451 (604)

5. Primary Outcome: The Number of Patients Reporting Any Treatment-emergent Adverse Event.
Description: To assess the safety and tolerability of visible fluorescent injectate (VFI)™ (employing the FAST PV Technology™) in chronic dialysis patients with extremely reduced or no renal function subjects will be monitored for adverse events and serious adverse events following administration of the first dose of the study drug through the end of the study.
  Treatment-emergent adverse events will be tabulated by system organ class, preferred term, and cohort. Treatment-emergent AEs will be further classified by severity and relationship to study product.
Time Frame: 59 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 10
Participants | 8

6. Primary Outcome: The Number of Patients Reporting Any Treatment-emergent Serious Adverse Event.
Description: as for outcome 5
Time Frame: 59 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 10
Participants | 3

7. Primary Outcome: The Number of Patients Reporting Any Drug-related Treatment-emergent Serious Adverse Event.
Description: as for outcome 5
Time Frame: 59 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 10
Participants | 0

8. Primary Outcome: The Number of Patients Reporting Any Drug Related Treatment-emergent Adverse Event.
Description: as for outcome 5
Time Frame: 59 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 10
Participants | 4

ADVERSE EVENTS:
Time Frame: Enrollment through Discharge, possibly up to 59 days.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1) — GI Bleed, not drug related.
Volume Overload (Vascular disorders) | 2 (2) — Not drug related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)
Viral Syndrome (Infections and infestations) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Clotted Fistula (General disorders) | 1 (1)
Fistula Pseudoaneurysm (General disorders) | 1 (1)
Volume Overload (Vascular disorders) | 1 (1)
Elevated CPK (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
One patient's PV and ISV were not evaluable post dialysis due to a sampling error.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04733664/Prot_000.pdf
  • Informed Consent Form (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04733664/ICF_001.pdf